CLINICAL TRIAL: NCT04088591
Title: High-dose Intravenous Vitamin C as an Adjunctive Treatment for Sepsis in Rwanda: a Feasibility Trial
Brief Title: High-dose Intravenous Vitamin C as an Adjunctive Treatment for Sepsis in Rwanda
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Recent studies suggest an increase in mortality due to high-does Vitamin C
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Rwanda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20018390
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Sepsis
Keywords: Sepsis; Shock, Septic; ascorbic acid;
MeSH Terms: conditions — Sepsis; Shock | interventions — Ascorbic Acid; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment arm (Experimental): The study drug is ascorbic acid is 200mg/kg/day divided over 4 doses per day and delivered in 50 ml of 5% dextrose in water intravenously over a total duration of 96 hours.
  Interventions: Drug: Ascorbic Acid 500Mg/Ml Inj
- Placebo arm (Placebo Comparator): The placebo is 50ml of 5% dextrose in water and will be administered 4 doses per day over a total duration of 96 hours
  Interventions: Drug: Dextrose in Water

INTERVENTIONS:
Drug: Ascorbic Acid 500Mg/Ml Inj — Ascorbic acid 200mg/kg/day administered upon suspicion or confirmation of sepsis every 6 hours for a total duration of 96 hours
  Arms: Treatment arm
Drug: Dextrose in Water — 50 ml of 5% dextrose in water every 6 hours for a total duration of 96 hours
  Arms: Placebo arm

SUMMARY:
This feasibility study serves to determine if it is possible to perform a powered randomized control trial of high-dose intravenous vitamin C (ascorbic acid) as an adjunctive medication in the management of sepsis and septic shock in Rwanda. Further data will be collected including Sequential Organ Failure Assessment (SOFA) score, Universal Vital Assessment (UVA) score, duration of vasopressors, mortality and other key indicators to possibly determine the impact of vitamin C on organ failure and clinical course. A total of 24 patients with a diagnosis of sepsis or septic shock will be recruited after obtaining informed consent at the University Teaching Hospital of Kigali (CHUK) and will be randomized in a 1:1 fashion to receive drug or placebo. Both treatment arms will receive standard treatment (intravenous fluids, antibiotics, vasopressors as needed, etc.) in addition to study drug or placebo.

During the course of the study, any difficulties encountered will be recorded and will inform process improvements for a full randomized control, if it is indeed considered possible to perform the definitive trial.

DETAILED DESCRIPTION:
General objectives:

This study will primarily determine if it is possible to perform a powered randomized control trial of the administration of intravenous high-dose vitamin C for the treatment of sepsis or septic shock in the tertiary care setting in Rwanda. Additionally, the study will also attempt to assess any impact vitamin C has on morbidity and mortality.

Specific objectives:

This feasibility study will determine the possibility of and any difficulties encountered with:

* Storage of vitamin C solution
* Obtaining informed consent
* Pharmaceutical preparation of vitamin C for intravenous administration
* Protection of Vitamin C solution from light during administration
* Nursing acquisition of vital signs during course of administration
* Acquisition of key labs
* Retrieval of data from patient chart for analysis

Hypothesis:

It is expected that the study will be feasible. We also believe that a difference indicating benefit will be seen when comparing the patients receiving the study drug compared to placebo in such key areas as hospital length of stay, duration of mechanical ventilation or vasopressors, and mortality.

Primary outcome:

The primary outcome of this study is the determination of the feasibility of performing a randomized control trial of high-dose intravenous vitamin C in the management of septic shock.

Methodology:

Institutional Review Board approval will be sought at he University of Rwanda College of Medicine and Health Sciences (UR CMHS), at the study site University Teaching Hospital of Kigali (CHUK), and at Virginia Commonwealth University. This feasibility study will be carried out in a double-blind randomized control trial format. The clinical trial will be registered with ClincalTrials.gov and with the Pan African Clinical Trial Registry (PACTR).

Adult patients admitted to the emergency department, medicine ward, surgery ward, obstetrics and gynecology ward, and intensive care unit (ICU) at CHUK will be screened by study personnel for possible inclusion on weekdays from 8:00 A.M. to 5:00 P.M. Patients will be screened for sepsis or septic shock with the following criteria to determine if they are eligible to participate in the study:

1. Presence of organ dysfunction brought on by sepsis. This defined by an increase of two or more points in the qSOFA score
2. Strong suspicion or confirmation of infection If a patient meets both of these criteria, informed consent will be sought from the patient-if the patient is not able to consent, consent will be obtained from family members of the patient (further details of informed consent addressed below).

If informed consent is obtained, the patient will receive either intravenous placebo or intravenous vitamin C. Placebo will be 50ml of 5% dextrose in water and will be administered 4 doses per day over a total duration of 96 hours. The study drug will be obtained from McGuff Pharmaceuticals (Santa Ana, California, USA) and will be intravenous vitamin C (ascorbic acid) 200mg/kg/day divided over 4 doses and delivered in 50 ml of 5% dextrose and water over a total duration of 96 hours. In order to properly store and prepare the study drug, assistance will be sought from pharmacy at CHUK and the manufacturer's instructions will be followed. Patients will be randomized in a 1:1 fashion to receive study drug or placebo using Research Randomizer. Both placebo and study drug will be administered in shrouding material to protect the ascorbic acid and to preserve blinding. The study drug will be administered within two to four hours of diagnosis of sepsis or septic shock.

Patients in both arms will receive the standard of care regarding intravenous fluid resuscitation, but the antibiotic regimen will be altered from the standard of care (but the regimen will be the same in both trial arms). The standard of care for sepsis and the standard of care in prior studies that assessed high-dose intravenous vitamin C in sepsis and septic shock is prompt infusion of broad-spectrum intravenous antibiotics and prompt infusion of intravenous fluids. Sepsis still tends to be treated with ceftriaxone (with or without metronidazole) at CHUK yet very high levels of resistance have been shown.15 Therefore, for patients who participate in this study, the empiric antibiotic will be meropenem (with or without anti-tuberculosis and antimalarial drugs if indicated) and pharmacy will coordinate with this study to ensure meropenem is available at all times. In the event a patient is unable to afford meropenem, this will be covered by the study (this has now been added to the budget). Regarding intravenous fluid resuscitation, in prior studies of high-dose intravenous ascorbic acid, prompt administration of high-volume intravenous normal saline was employed; however, it has been shown that this mode of fluid resuscitation results in a greater mortality compared to standard of care in a randomized controlled trial in sub-Saharan Africa reported in the Journal of the American Medical Association in 2017.16 Therefore, the standard of care in terms of intravenous fluid resuscitation in Rwanda will not be altered.

Prior to administration of the vitamin C, the patient's blood will be drawn and collected in order to assess the following values: creatinine, total bilirubin, white blood cell count, platelet count, PaO2, lactate, and ascorbic acid level and these labs will be drawn at 24, 48, 72, and 96 hours, with the exception of plasma ascorbic acid level, which will be drawn at enrollment and at 24 hours. Glasgow Coma Scale score, respiratory rate, and blood pressure will be measured at enrollment and at 24, 48, 72, and 96 hours. When a patient with diabetes is enrolled, venous samples must be drawn to assess glucose levels-fingerstick blood glucose levels have been shown to be not accurate for patient with hyperglycemia. Of note, neither the patients nor their family members will be responsible for payment for the laboratory assays and these will all be funded by this study.

The safety profile of high-dose ascorbic acid has been well verified and side effects have been shown to be minimal. A metanalysis of five clinical trials of high-dose intravenous vitamin C, which included the studies performed by Fowler et al. and Zabet et al. demonstrated that no adverse reactions occurred in the 76 patients who received high-dose intravenous vitamin C. In the study performed by Nathans et al., 301 patients received high-dose intravenous vitamin C and no adverse events were reported.

The ascorbic acid package insert from McGuff Pharmaceuticals indicates that possible adverse reactions include oxalate nephropathy, hemolysis in patients with glucose-6-phosphate dehydrogenase deficiency, and pain and swelling at the infusion site.

While there is a theoretical risk of hyperoxaluria and oxalate nephropathy, this has not been seen in clinical trials of high-dose intravenous vitamin C; yet, patients with a history of kidney stones will be excluded. The study participant will have his/her renal function monitored daily during the study period. Patients with a known history of glucose-6-phosphatase-dehydrogenase (G6PD) deficiency will be excluded and every patient will have his/her hemoglobin measured daily. Patients will be monitored for pain and swelling at the infusion site and if this occurs the infusion will be stopped, a cold compress will be applied, and the infusion will be restarted at 50% of the prior rate.

While it is not likely that an adverse reaction will occur, in the event an adverse reaction occurs, the study recruiter/coordinator will stop the infusion, notify the PI immediately, and complete an incident report form (included in the IRB application packet) will be completed. The incident report sheet will be available in all clinical care areas where the patient may receive intravenous high-dose ascorbic acid (e.g., internal medicine ward, intensive care unit, etc.). If the adverse event occurs outside the study recruiter/coordinator's work hours, the in-charge nurse will perform these duties. The UR-CMHS IRB and other IRBs will be notified of the event as well.

Study site:

University Teaching Hospital of Kigali (CHUK)

Study design:

Feasibility double-blind randomized control trial

Data collection:

Key metrics as per above, including SOFA and UVA scores and laboratory values, will be recorded in the patient's chart by nursing or study personnel and will be entered into REDCap (a secure web-based application for storage and management of data) at the time of patient discharge or death.

Study period:

The study will be conducted from November 2019 until 24 patients have been recruited and complete the study-it is expected that the study will conclude in November 2020.

Sample size:

The sample size will be 24 patients, with 12 patients in the treatment arm of the trial and 12 patients in the placebo arm.

Ethical considerations:

Informed consent:

Patients or surrogate decision maker (in the event of patient's incapacity to make decisions and provide consent, in most circumstances family members) will be fully informed of all risks and benefits of participating in the trial. Risk of intravenous high-dose vitamin C have been shown to be minimal. The decision maker will be informed that the patient may receive placebo or study drug. The informed consent form will be available in both English and Kinyarwanda and if the decision maker is illiterate the form will be read to him or her. All questions will be answered in full.

Confidentiality measures:

During the study we will make sure that the privacy and confidentiality of participants are respected. All research team members will avoid discussing sensitive information concerning individuals where they may be overheard or leave individual's information, either on paper or on computer screens, where they can be seen by other patients/subjects, unauthorized health care staff or the public.

Regarding data collection and storage, the investigator will create a dataset key and assign a unique identifier to each patient selected for chart review for recording individual patient study data. Resultant study data will therefore be de-identified and will then be stored electronically in password protected files on an encrypted computer. The PI will be responsible for overseeing data management.

Data will be accessible only by the research team, overseen by the Principal Investigator, who will possess passwords and keys to enter. Only de-identified data untraceable to study participants will be retained after study completion by the study investigators.

Subsequently, only the named study investigators will have access to the de-identified data. De-identified data may be shared with the health facility leadership and regulatory bodies as may be required for oversight.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 18 and 80 who provide informed consent (or consent obtained by family member if patient is incapacitated) AND
* Patients with a strong suspicion or confirmation of infection AND
* Presence of organ dysfunction brought on by sepsis. This defined by an increase of two or more points in the qSOFA score

Exclusion Criteria:

* Known allergic reaction to ascorbic acid
* Pregnant patients or those who may be pregnant
* History of renal stones
* History of end-stage renal disease (ESRD) requiring dialysis
* History of glucose-6-phosphatase dehydrogenase (G6PD) deficiency
* History of hemochromatosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility - number of participants recruited | 12 months
  Recruitment feasibility will be measured using the number of participants enrolled over a one-year period
Feasibility - number of participants adherence to study protocol | 96 hours
  Study protocol feasibility will be measured using the number of participants on whom all vital signs, labs, and placebo / trial drug administration is fully adhered to in a 96-hour period

SECONDARY OUTCOMES:
Change in SOFA score | 4 days
  SOFA is a single score based on patient status on six different biological systems: respiratory, cardiovascular, hepatic, coagulation, renal, and neurological. Scores range from 0 to 24 with higher scores indicated worse status. A greater reduction in mean SOFA score is expected in treatment arm compared to placebo arm.
Change in Universal Vital Assessment (UVA) score | 4 days
  UVA is a single score based on patient temperature, heart and respiratory rates, systolic blood pressure, oxygen saturation, Glasgow coma scale score and HIV serostatus A greater reduction in mean UVA score is expected in treatment arm compared to placebo arm.
Rate of acute kidney injury | 7 days
  Proportion of patients developing acute kidney injury will be lower in treatment arm compared to placebo arm
Rate of thrombocytopenia | 7 days
  Proportion of patients developing thrombocytopenia (platelet count less than 150,000 / uL) will be lower in treatment arm compared to placebo arm
Rate of mechanical ventilation | 7 days
  Proportion of patients receiving mechanical ventilation will be lower in treatment arm compared to placebo arm
Duration of mechanical ventilation | 7 days
  Mean duration of mechanical ventilation when used will be lower in treatment arm compared to placebo arm
Rate of vasopressor usage | 7 days
  Proportion of patients receiving vasopressor will be lower in treatment arm compared to placebo arm
Duration of vasopressor usage | 7 days
  Mean duration of vasopressor when used will be lower in treatment arm compared to placebo arm
Rate of acute respiratory distress syndrome | 7 days
  Proportion of patients developing acute respiratory distress syndrome will be lower in treatment arm compared to placebo arm
Length of intensive care unit stay | 30 days
  Mean length of stay in intensive care unit will be shorter in treatment arm compared to placebo arm
Length of hospital stay | 30 days
  Mean length of stay in hospital will be shorter in treatment arm compared to placebo arm
Rate of in-hospital mortality | 30 days
  Mortality rate will be lower in treatment arm compared to placebo arm

CONTACTS AND LOCATIONS:
Overall Officials: Dennis A Hopkinson, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- University Teaching Hospital of Kigali, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data will be shared, after de-identification, to researchers who present to the authors a methodologically sound proposal for meta-analysis. Proposals should be directed to dahopk@gmail.com.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 5 years after study publication.
Access Criteria: This data will be made available to researchers who present to the authors a methodologically sound proposal for meta-analysis.